CLINICAL TRIAL: NCT00002496
Title: PHASE III TRIAL TO PRESERVE THE LARYNX: INDUCTION CHEMOTHERAPY AND RADIATION THERAPY VERSUS CONCOMITANT CHEMOTHERAPY AND RADIATION THERAPY VERSUS RADIATION THERAPY
Brief Title: Radiation Therapy With or Without Chemotherapy in Treating Patients With Advanced Cancer of the Larynx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RTOG-9111; CDR0000077756; EST-R9111; SWOG-9201
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Drug Therapy; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: chemotherapy
Drug: cisplatin
Drug: fluorouracil
Procedure: conventional surgery
Radiation: low-LET cobalt-60 gamma ray therapy
Radiation: low-LET electron therapy
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known if chemotherapy plus radiation therapy is more effective than radiation therapy alone in treating patients with advanced cancer of the larynx.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without chemotherapy in treating patients with advanced cancer of the larynx.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare, in a phase III setting, overall and disease-free survival with preservation of laryngeal function in patients with stage III/IV squamous cell carcinoma of the glottic and supraglottic larynx treated with cisplatin/fluorouracil (CDDP/5-FU) followed by radiotherapy vs. concomitant radiotherapy plus CDDP vs. radiotherapy alone. II. Compare the tumor response after completion of chemotherapy but prior to initiation of radiotherapy with that following completion of radiotherapy and concurrent chemotherapy. III. Compare the patterns of relapse (local and regional recurrence and distant metastasis) with these treatments. IV. Compare the incidence of second primary tumors in patients treated on these three regimens. V. Compare the acute and chronic adverse effects of these three regimens. VI. Compare the morbidity experienced with neck dissection and/or laryngeal salvage surgery following treatment with these regimens. VII. Compare quality of life of patients with laryngeal preservation vs. patients requiring salvage laryngectomies. VIII. Compare the quality of life of patients receiving radiotherapy alone vs. those receiving chemotherapy as well.

OUTLINE: Randomized study. Patients on any arm, clinically staged N+ undergo neck dissection following completion of radiotherapy. Arm I: 2-Drug Combination Chemotherapy followed by Radiotherapy. Cisplatin, CDDP, NSC-119875; Fluorouracil, 5-FU, NSC-19893; followed by regional irradiation using linear accelerators with photon energies of 1.25-6 MV, electron energies of 8-17 MeV, or Co60. Arm II: Radiotherapy plus Single-Agent Chemotherapy/Radiosensitization. Regional irradiation using equipment as in Arm I; plus CDDP. Arm III: Radiotherapy. Regional irradiation using equipment as in Arm I.

PROJECTED ACCRUAL: 546 patients (182/arm) will be entered over approximately 3 years. If any arm is clearly inferior in laryngectomy-free survival after 137 patients have completed 2 years of follow-up study, that arm will be closed to further accrual. A second interim analysis will be conducted after 410 patients have completed 2 years of follow-up.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy-proven, previously untreated, squamous cell carcinoma of the glottic and supraglottic larynx that would normally require total laryngectomy Stage III/IV disease (excluding T1 and M1) Endoscopic tumor staging required within 4 weeks of entry Tumors must be considered resectable and potentially curable with conventional surgery and radiotherapy T4 disease limited to: Up to 1 cm invasion of the base of tongue Questionable cartilage invasion on CT (clinically T3) Measurable disease required No synchronous primary tumors No subglottic tumors

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60%-100% Hematopoietic: (obtained within 3 weeks of entry) WBC at least 3,500 Platelets at least 100,000 Hepatic: Not specified Renal: (obtained within 2 weeks of entry) Creatinine clearance at least 50 mL/min (measured or calculated) Serum calcium normal Cardiovascular: Status adequate to tolerate all protocol therapy Pulmonary: Status adequate to tolerate all protocol therapy Other: Nutritional status adequate to tolerate all protocol therapy Mental status adequate to follow instructions and keep appointments No second malignancy except nonmelanomatous skin cancer (Patients who have been disease-free for at least 3 years following treatment for a prior cancer may be eligible at the discretion of the protocol chairman) Negative pregnancy test required of fertile women Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior therapy Chemotherapy: No prior therapy Endocrine therapy: No prior therapy Radiotherapy: No prior radiotherapy to the head and neck Surgery: No prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-08; Primary Completion 2002-08 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helmuth Goepfert, MD, Study Chair — M.D. Anderson Cancer Center; George L. Adams, MD, Study Chair — Masonic Cancer Center, University of Minnesota; David E. Schuller, MD, Study Chair — Ohio State University Comprehensive Cancer Center
Locations (18):
- United States (17):
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Ireland Cancer Center, Cleveland, Ohio
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Background] Dilling TJ, Bae K, Paulus R, Watkins-Bruner D, Garden AS, Forastiere A, Kian Ang K, Movsas B. Impact of gender, partner status, and race on locoregional failure and overall survival in head and neck cancer patients in three radiation therapy oncology group trials. Int J Radiat Oncol Biol Phys. 2011 Nov 1;81(3):e101-9. doi: 10.1016/j.ijrobp.2011.01.013. Epub 2011 May 5. PMID 21549515
- [Background] Coyne JC, Pajak TF, Harris J, Konski A, Movsas B, Ang K, Watkins Bruner D; Radiation Therapy Oncology Group. Emotional well-being does not predict survival in head and neck cancer patients: a Radiation Therapy Oncology Group study. Cancer. 2007 Dec 1;110(11):2568-75. doi: 10.1002/cncr.23080. PMID 17955501
- [Background] Machtay M, Moughan J, Trotti A, Garden AS, Weber RS, Cooper JS, Forastiere A, Ang KK. Factors associated with severe late toxicity after concurrent chemoradiation for locally advanced head and neck cancer: an RTOG analysis. J Clin Oncol. 2008 Jul 20;26(21):3582-9. doi: 10.1200/JCO.2007.14.8841. Epub 2008 Jun 16. PMID 18559875
- [Background] Siddiqui F, Pajak TF, Watkins-Bruner D, Konski AA, Coyne JC, Gwede CK, Garden AS, Spencer SA, Jones C, Movsas B. Pretreatment quality of life predicts for locoregional control in head and neck cancer patients: a radiation therapy oncology group analysis. Int J Radiat Oncol Biol Phys. 2008 Feb 1;70(2):353-60. doi: 10.1016/j.ijrobp.2007.06.024. Epub 2007 Sep 24. PMID 17889449
- [Background] Spiegel D, Kraemer HC. Emotional well-being does not predict survival in head and neck cancer patients: a Radiation Therapy Oncology Group study. Cancer. 2008 May 15;112(10):2326-7; author reply 2327-8. doi: 10.1002/cncr.23435. No abstract available. PMID 18338746
- [Background] Konski A, Bhargavan M, Owen J, et al.: The price of failure: economic analysis of recurrence and complications of patients treated on RTOG 91-11. [Abstract] The American Radium Society 89th Annual Meeting, May 5-29, 2007, Amsterdam, Netherlands. A-SS-6, 3, 2007.
- [Background] O'Meara EA, Machtay M, Moughan J, et al.: Associations between radiation doses to pharyngeal regions and severe late toxicity in head and neck cancer patients treated with concurrent chemoradiotherapy: an RTOG analysis. [Abstract] Int J Radiat Oncol Biol Phys 69 (3): A-96, S54-5, 2007.
- [Background] Konski AA, Bhargavan M, Owen J, et al.: The addition of chemotherapy to radiation is cost-effective in the treatment of patients with locally advanced laryngeal cancer: an economic analysis of Radiation Therapy Oncology Group (RTOG) 91-11. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-115, S66, 2006.
- [Background] Machtay M, Moughan J, Trotti A, et al.: Pre-treatment and treatment related risk factors for severe late toxicity after chemo-RT for head and neck cancer: an RTOG analysis. [Abstract] J Clin Oncol 24 (Suppl 18): A-5500, 280s, 2006.
- [Background] Mukherji SK, Toledano AY, Beldon C, Schmalfuss IM, Cooper JS, Sicks JD, Amdur R, Sailer S, Loevner LA, Kousouboris P, Ang K. Interobserver reliability of computed tomography-derived primary tumor volume measurement in patients with supraglottic carcinoma. Cancer. 2005 Jun 15;103(12):2616-22. doi: 10.1002/cncr.21072. PMID 15887218
- [Background] Bourhis J, Amand C, Pignon JP, et al.: Update of MACH-NC (Meta-Analysis of Chemotherapy In Head & Neck Cancer ) database focused on concomitant chemotherapy. [Abstract] J Clin Oncol 12 (Suppl 14): A-5505, 489s, 2004.
- [Background] Konski AA, Pajak T, Movsas B, et al.: Socio-demographic variables influence outcome in Radiation Therapy Oncology Group head and neck trials. [Abstract] Proceedings of the American Society of Clinical Oncology 22 (Suppl 14): A-6043, 529s, 2004.
- [Background] Movsas B, Konski A, Pajak T, et al.: Quality of life (QOL) variables influence local regional control in Radiation Therapy Oncology Group (RTOG) headsneck trials (9003 and 9111). [Abstract] Int J Radiat Oncol Biol Phys 60 (1 Suppl 1): A-199, S252, 2004.
- [Result] Forastiere AA, Maor M, Weber RS, et al.: Long-term results of intergroup RTOG 91-11: a phase III trial to preserve the larynx--Induction cisplatin/5-FU and radiation therapy versus concurrent cisplatin and radiation therapy versus radiation therapy. [Abstract] J Clin Oncol 24 (Suppl 18): A-5517, 284s, 2006.
- [Result] Forastiere AA, Goepfert H, Maor M, Pajak TF, Weber R, Morrison W, Glisson B, Trotti A, Ridge JA, Chao C, Peters G, Lee DJ, Leaf A, Ensley J, Cooper J. Concurrent chemotherapy and radiotherapy for organ preservation in advanced laryngeal cancer. N Engl J Med. 2003 Nov 27;349(22):2091-8. doi: 10.1056/NEJMoa031317. PMID 14645636
- [Result] Weber RS, Berkey BA, Forastiere A, Cooper J, Maor M, Goepfert H, Morrison W, Glisson B, Trotti A, Ridge JA, Chao KS, Peters G, Lee DJ, Leaf A, Ensley J. Outcome of salvage total laryngectomy following organ preservation therapy: the Radiation Therapy Oncology Group trial 91-11. Arch Otolaryngol Head Neck Surg. 2003 Jan;129(1):44-9. doi: 10.1001/archotol.129.1.44. PMID 12525193
- [Result] Maor MH, Berkey B, Forastiere A, et al.: Larynx preservation and tumor control in stage III and IV laryngeal cancer: a three-arm randomized intergroup trial: RTOG 91-11. [Abstract] Int J Radiat Oncol Biol Phys 54(2 suppl 1): 2-3, 2002.
- [Result] Wolf GT. Commentary: phase III trial to preserve the larynx: induction chemotherapy and radiotherapy versus concurrent chemotherapy and radiotherapy versus radiotherapy--intergroup trial R91-11. J Clin Oncol. 2001 Sep 15;19(18 Suppl):28S-31S. No abstract available. PMID 11560968